CLINICAL TRIAL: NCT04927858
Title: Prevalence of Cardiovascular Disease in Swedish Patients With Type 2 Diabetes and in Patients Initiating on Empagliflozin
Brief Title: A Study Using Swedish Registries to Find Out How Many People With Type 2 Diabetes Had Cardiovascular Disease and Started Treatment With Empagliflozin Between 2015 and 2017
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0190
Record Dates: First submitted 2021-06-10; First posted 2021-06-16 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population 1: Patients ≥ 18 years old on 31st of December 2017 with Type 2 Diabetes Mellitus (T2DM) who were alive on 31st of December 2017 and had at least one registration in the Swedish National Diabetes Registry (NDR) between 1996 - 2017.
- Population 2: Population 2 is a sub-population of population 1. Patients with Type 2 Diabetes Mellitus (T2DM) who were initiated on Empagliflozin between 1st of January 2015 and 31st of December 2017, who had at least one registration in the Swedish National Diabetes Register (NDR).
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin
  Groups: Population 2

SUMMARY:
This study aims to describe the prevalence of type 2 diabetes mellitus (T2DM) patients with established cardiovascular disease (CVD) according to the (Empagliflozin) Cardiovascular Outcome Event Trial in Type 2 Diabetes Mellitus Patients (EMPA-REG OUTCOME (ERO)) study definition in a Swedish population.

The aim was also to describe the prevalence of established CVD according to ERO study definition in patients with T2DM who initiates treatment with empagliflozin

ELIGIBILITY:
Inclusion criteria

Population 1: 'Prevalence of a history of cardiovascular disease (CVD) among persons with type 2 diabetes mellitus (T2DM) who were alive on 31 December 2017' :

* Diagnosed with T2DM in Sweden
* Alive on 31 December 2017
* At least one registration in the Swedish National Diabetes Register (NDR)
* Each patient provides informed consent for inclusion in the register

Population 2: 'Prevalence of a history of CVD among persons with type 2 diabetes who started empagliflozin treatment between 1 January 2015 and 31 December 2017':

* Diagnosed with T2DM in Sweden
* Alive on 31 December 2017
* Initiated on empagliflozin between 1 January 2015 and 31 December 2017
* At least one registration in the NDR
* Each patient provides informed consent for inclusion in the register

Exclusion criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with T2DM and age ≥18 years on 2017-12-31 and who had at least one registration in the Swedish National Diabetes Register (NDR) between 1996 - 2017.
Sampling Method: Non-Probability Sample
Enrollment: 460558 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim AB, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets
Supporting Information: SAP, CSR
Time Frame: After all regulatory activities are completed in the US and European Union (EU) for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This retrospective study assessed the prevalence of cardiovascular disease in Swedish patients with type 2 diabetes mellitus (T2DM) and in Swedish patients with T2DM initiating on empagliflozin.
Pre-assignment Details: This study was conducted using data collected from the Swedish National Diabetes Register (NDR) as well as the Swedish Prescribed Drug Register (SPDR) and the Swedish National Patient Register (NPR) (National Board of Health and Welfare). The observation period was from 1996 to end of December 2017.
Groups:
- Overall Type 2 Diabetes Mellitus Population: This arm included all patients ≥ 18 years old on 31st of December 2017 with Type 2 Diabetes Mellitus (T2DM) who were alive on 31st of December 2017 and had at least one registration in the Swedish National Diabetes Registry (NDR) between 1996 - 2017.
Period: Overall Study
Arm/Group | Overall Type 2 Diabetes Mellitus Population
Started | 460558
Treated With Empagliflozin (Patients with Type 2 Diabetes Mellitus (T2DM) who were initiated on Empagliflozin between 1st of January 2015 and 31st of December 2017, who had at least one registration in the Swedish National Diabetes Register (NDR).) | 16985
Completed | 460558
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients ≥ 18 years old on 31st of December 2017 with Type 2 Diabetes Mellitus (T2DM) who were alive on 31st of December 2017 and had at least one registration in the Swedish National Diabetes Registry (NDR) between 1996 - 2017.
Arm/Group | Overall Type 2 Diabetes Mellitus Population
Number analyzed (Participants) | 460558
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197459
  Male | 263099
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of a History of Cardiovascular Disease (CVD) Among Swedish Patients With Type 2 Diabetes Mellitus (T2DM) Who Were Alive on 31st of December 2017
Description: The number of participants with a history of CVD and without a history of CVD among patients who had Type 2 Diabetes Mellitus (T2DM) and were ≥ 18 years old on 31st of December 2017, and were alive on 31st of December 2017, and had at least one registration in the Swedish National Diabetes Registry (NDR) between 1996 - 2017 is reported. History of CVD was defined as a history of either coronary heart disease, stroke, amputation, percutaneous coronary intervention, coronary artery bypass surgery, peripheral vascular disease, or carotid or femoral angioplasty.
Time Frame: Data collected at the index date 31st of December 2017, data covering a time period from 1996 until 2017, up to 21 years.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Type 2 Diabetes Mellitus Population
Number analyzed (Participants) | 460558
Participants
  With history of CVD | 130508
  Without history of CVD | 330050

2. Primary Outcome: Prevalence of a History of CVD Among Swedish Patients With T2DM Who Started Empagliflozin Treatment Between 1st of January 2015 and 31st of December 2017
Description: The number of participants with a history of CVD and without a history of CVD among patients with Type 2 Diabetes Mellitus (T2DM) who were initiated on Empagliflozin between 1st of January 2015 and 31st of December 2017, who had at least one registration in the Swedish National Diabetes Register (NDR). History of CVD was defined as a history of either coronary heart disease, stroke, amputation, percutaneous coronary intervention, coronary artery bypass surgery, peripheral vascular disease, or carotid or femoral angioplasty.
Time Frame: as for outcome 1
Population: All patients with Type 2 Diabetes Mellitus (T2DM) who were initiated on Empagliflozin between 1st of January 2015 to 31st of December 2017, who had at least one registration in the Swedish National Diabetes Register (NDR).
Measure: Count of Participants; unit: Participants
Groups:
- Empagliflozin Type 2 Diabetes Mellitus Population: Patients with Type 2 Diabetes Mellitus (T2DM) who were initiated on Empagliflozin between 1st of January 2015 and 31st of December 2017, who had at least one registration in the Swedish National Diabetes Register (NDR).
Arm/Group | Empagliflozin Type 2 Diabetes Mellitus Population
Number analyzed (Participants) | 16985
Participants
  With history of CVD | 1952
  Without history of CVD | 15033

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: As this is a non-interventional study with secondary use of data retrieved from Swedish Databases safety monitoring and safety reporting on an individual case level is not applicable. All-Cause Mortality, Serious Adverse Events and Other Adverse Events are not collected in the database. "0" total Number of Participants at Risk means "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed".
Arm/Group | Overall Type 2 Diabetes Mellitus Population
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT04927858/Prot_SAP_001.pdf